CLINICAL TRIAL: NCT00502749
Title: Feasibility, Safety, and Effect of an Exercise Program for Adolescents and Young Adults With Cancer
Brief Title: Exercise Program for Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ID02-329
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; Exercise; Quality of Life; Questionnaire; Survey
MeSH Terms: conditions — Leukemia; Lymphoma; Motor Activity | interventions — Resistance Training; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise program (Experimental): Daily (Monday-Friday) 45-minute group physical exercise program during each hospital admission for three months or individual 20 minute session bedside.
  Interventions: Behavioral: Exercise program; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Exercise program — Daily group or personal exercise programs designed to promote flexibility, endurance, and strength.
Behavioral: Questionnaires — Questionnaires taking 15 minutes to complete.
  Other Names: Survey

SUMMARY:
This pilot study will examine the safety, feasibility, and effect on quality of life of moderate physical activity on adolescent and young adult patients who are admitted to the hospital periodically for routine chemotherapy. Patients will be asked to participate in daily physical exercise during hospital admissions over a three-month period. Exercise sessions will be monitored and guided by M.D. Anderson physical therapists, a personal trainer, and Dr. Michael Rytting, pediatric oncologist. The personal trainer will meet with each participant for reinforcement and to provide an opportunity for exercise between hospitalizations. If results are positive, the study will be extended to a larger cohort of patients.

DETAILED DESCRIPTION:
Patients who are staying at M.D. Anderson for inpatient chemotherapy treatment will take part in this study.

Participants in this study will be asked to take part in either mild physical exercise by themselves for 20 minutes a day, or group exercise sessions of moderate intensity once a day. Each participant will be evaluated by a physical therapist before participation.

Exercise programs will be designed for each individual. Participants will be encouraged to attend group sessions and continue the exercise program during the time they are outpatients. Participants will also have the opportunity to work with a personal trainer.

The group exercise program takes from 45 minutes to one hour, and will be performed under the guidance of certified physical therapists and a personal trainer in the Pedi-Dome located on the ninth floor of the Alkek Tower of M.D. Anderson. Participants who are not feeling well enough to come to the Pedi-Dome on a given day will have the opportunity to exercise in their hospital rooms with a physical therapist or trainer for 20 minutes.

The exercises are designed to promote flexibility, endurance, and strength. They include activities such as stretching, pilates-yoga, aerobics, step aerobic training, use of stationery bikes, and the use of therapeutic exercise balls, cuff weights, and dumbbells. The activities will be tailored to each individual's abilities and special needs.

The total length of participation in this study is three months. Participants will be asked to exercise each day that they are an inpatient and well enough to participate. Participants will be encouraged to continue exercise and participation in the exercise program when they are outpatients, but it will not be required. Participants will fill out short questionnaires and be evaluated for quality of life, fatigue, physical strength, and medical and nutritional status four times: at the time of enrollment in the study, and at one, two, and three months after enrollment. The questionnaires will take about 15 minutes to complete.

This is an investigational study. A total of 40 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents and young adults with leukemia/lymphoma between the ages of 12 and 25 years old.
2. Leukemia/lymphoma patients admitted for chemotherapy with an anticipated hospital stay of at least three days.

Exclusion Criteria:

1. Patients with an underlying condition that precludes moderate exercise due to safety.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2003-02; Primary Completion 2007-11 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Exercise Participation Rate | Baseline to 3 months
  Participation in exercise program as measured through group attendance examined from study entry to three months later. Exercise participation rate was examined across 4 timepoints corresponding to inpatient chemotherapy treatments, and calculated as number of those exercising in each period divided by total participants in that period.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Askins, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org